CLINICAL TRIAL: NCT07084181
Title: Get Your Rear In Gear Study: Feasibility of Using Fitness Tracker to Assess Activity Level and Toxicities in Patients With Localized/Advanced Colorectal Cancer: A Fox Chase Cancer Center Pilot Study
Brief Title: Fitbit Assessed PS in Colorectal Cancer
Status: Completed | Type: Observational
Sponsor: Fox Chase Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 16-8023; 16-8023 (Other: Fox Chase Cancer Center)
Record Dates: First submitted 2025-07-16; First posted 2025-07-24 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Colorectal Cancer (Diagnosis)
Keywords: Colorectal Cancer; Patient Reported Outcomes; Fitness Tracker
MeSH Terms: conditions — Colorectal Neoplasms; Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and serum frozen and stored
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Primary Objective

To assess the feasibility of activity tracking using Fitbit device in terms of compliance (defined as at least 75% of patients complying with instructions to wear the device, for at least 12 hours a day on at least 3 of the 4 assigned days) in patients undergoing therapy for localized and advanced colorectal cancer.

Secondary Objectives

* To determine if physician-assessed performance status correlates with FitbitTM assessed physical activity (using active-minutes data).
* To correlate baseline physical activity level as assessed by FitbitTM with incidence of grade III or higher toxicities experienced during treatment
* To assess correlation between patient reported treatment related toxicities (PRO-CTCAE) and objective physical activity as measured by FitbitTM in patients treated for localized or metastatic cancers treated with chemotherapy
* To correlate baseline and interval change in physical activity levels as assessed by FitbitTM with post-surgical outcomes including inpatient length of stay, perioperative complications, post-operative 30-day mortality, and time to adjuvant treatment initiation (in days)

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Have histologically confirmed colorectal adenocarcinoma (Stage II-IV)
* Have an estimated life expectancy of greater than 3 months
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
* Should meet the following treatment arms:

  * Planned to undergo curative resection with or without neoadjuvant/adjuvant therapy for colorectal cancer (surgical arm);
  * Planned to undergo/undergoing systemic chemotherapy for localized/metastatic colorectal cancer - medical arm (patient enrolled on one arm may not enroll onto the other arm)
* Able to participate in some degree of physical activity (i.e. walking)
* Are undergoing treatment for their cancer at FCCC
* Ability to understand and willingness to sign a written informed consent and HIPAA consent

Exclusion Criteria:

* Inability to communicate in English.
* Already using a personal activity tracker
* Enrolled in another study in which physical activity is part or all of the therapeutic intervention or is being evaluated
* Pre-existing toxicity >grade II
* PS >3 for any reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — No concern
Study Population: Patients with colorectal cancer undergoing chemotherapy
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2017-02-15 (Actual); Primary Completion 2019-07-22 (Actual); Study Completion 2019-07-22 (Actual)

PRIMARY OUTCOMES:
Rate of usage | 4 days
  To assess the feasibility of activity tracking using Fitbit device in terms of compliance (defined as at least 75% of patients complying with instructions to wear the device, for at least 12 hours a day on at least 3 of the 4 assigned days) in patients undergoing therapy for localized and advanced colorectal cancer.
Steps | enrollment to 7 days
  tracker assessed step count

CONTACTS AND LOCATIONS:
Locations (1):
- Fox Chase Cancer Center, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
At reasonable request to PI
Supporting Information: Study Protocol, SAP, ICF, CSR

REFERENCES:
- [Background] Ward WH, Meeker CR, Handorf E, Hill MV, Einarson M, Alpaugh RK, Holden TL, Astsaturov I, Denlinger CS, Hall MJ, Reddy SS, Sigurdson ER, Dotan E, Zibelman M, Meyer JE, Farma JM, Vijayvergia N. Feasibility of Fitness Tracker Usage to Assess Activity Level and Toxicities in Patients With Colorectal Cancer. JCO Clin Cancer Inform. 2021 Jan;5:125-133. doi: 10.1200/CCI.20.00117. PMID 33492994